CLINICAL TRIAL: NCT04118218
Title: Determination of Predictive Clinical Signs of Effective Rhizolysis Using the DFL Questionnaire (Diagnosis of Facet Joint Origin Lumbago).
Brief Title: Determination of Predictive Clinical Signs of Effective Rhizolysis Using the DFL Questionnaire.
Acronym: Rhizolyse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: Dr BARAT (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-A01283-50
Record Dates: First submitted 2019-10-04; First posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-09

CONDITIONS: Rhizolysis; Diagnosis of Facet Joint Origin Lumbago
Keywords: DLF Questionnaire; rhizolysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Rhizolysis pain analysis — Definition of the subgroup of good clinical outcome after rhizolysis (called "effective" rhizolysis) by lumbar VAS or lower extremity pain VAS or Oswestry index decreased at 6 weeks after rhizolysis.
  The "efficiency" criterion based on the decrease in the dolorimeter or the Oswestry index corresponds to a decrease of at least 50% [1, 2, 3, 4].

SUMMARY:
Rhizolysis or lumbar thermocoagulation is a therapeutic proposal for certain types of chronic lower back pain that is resistant to medical treatment and outside the field of surgical indications.

A previous study has selected functional and physical signs selected by analysts and a group of experts from the modified "Delphi" prediction method. This study resulted in the creation of a questionnaire (DFL questionnaire) with 16 symptoms: 7 functional and 9 physical.

The aim of this new study is to select the symptoms that have the best positive predictive value among the 16 symptoms, to predict a good result of rhizolysis, on the criterion of their mitigation or disappearance in case of effective rhizolysis.

DETAILED DESCRIPTION:
The frequency of chronic lower back pain is a major economic and social problem. Indeed, there are numerous solutions that can be offered to patients, but sometimes they are unsatisfactory as medical treatments are often insufficiently effective, surgical techniques are often invasive and indications can be limited.

Rhizolysis or lumbar thermocoagulation is a therapeutic proposal for certain types of chronic lower back pain that is resistant to medical treatment and outside the field of surgical indications. This technique, which is minimally invasive, is low-risk for patients and is widely used. However, few studies have shown its effectiveness, so the level of evidence is not enough to make this technique accepted as a standard.

A previous study has selected functional and physical signs for joint involvement in lower back pain. This selection was made by analysts and a group of experts from the modified "Delphi" prediction method. This study resulted in the creation of a questionnaire (DFL questionnaire) with 16 symptoms: 7 functional and 9 physical.

The aim of this new study is to select the symptoms that have the best positive predictive value among the 16 symptoms, to predict a good result of rhizolysis, on the criterion of their mitigation or disappearance in case of effective rhizolysis.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from chronic lower back pain developing for more than 6 months and resistant to the medical treatments.
* Patients with an indication of lumbar rhizolysis for their chronic lower back pain with a facet component, the starting point of which corresponds to the L4L5 and/or L5S1 stages.
* Patient not objecting to their participation in the study.
* Subject registered with a social security scheme

Exclusion Criteria:

* Adults under judicial protection
* Adult under guardianship or trusteeship
* Pregnant women
* Minors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-12-12 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Predictive DFL symptoms | 6 weeks
  • Comparison of the "effective rhizolysis" and "non-effective rhizolysis" subgroups at 6 weeks postoperatively to select the symptoms with the highest positive predictive value among the 16 symptoms of the DFL questionnaire based on the criterion of effectiveness of a decrease of 50% of VAS or Oswestry

CONTACTS AND LOCATIONS:
Locations (1):
- Clairval Private Hospital, Marseille, PACA, France